CLINICAL TRIAL: NCT03220438
Title: Testing TMS Enhancement of Visual Plasticity in Schizophrenia
Brief Title: TMS Enhancement of Visual Plasticity in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator took another position elsewhere
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Laura Rowland, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HP-00072640
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMS (Active Comparator): rTMS
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham TMS (Sham Comparator): A sham coil will be used. This condition controls for the auditory artifacts induced by rTMS.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation

SUMMARY:
The major goal is to determine if Transcranial magnetic stimulation (TMS) enhances visual plasticity in schizophrenia. TMS sessions (sham/placebo and real TMS) will be conducted before two MRI scans with two weeks in-between to assess whether TMS stimulation to the visual cortex will enhance visual plasticity in patients with schizophrenia-spectrum disorders. This project may provide a better understanding of the underlying neurobiological mechanisms responsible for learning and memory deficits in schizophrenia.

DETAILED DESCRIPTION:
Learning and memory impairments are commonly observed in schizophrenia spectrum disorders. Alterations in "long-term potentiation" (LTP), a basic mechanism underlying learning and memory, may explain this impairment. This project will assess fMRI visual plasticity, thought to reflect LTP, in participants with and without schizophrenia spectrum disorders. Previous studies have shown that visual plasticity is impaired in schizophrenia. The major goal is to determine if Transcranial magnetic stimulation (TMS) enhances visual plasticity in schizophrenia. Transcranial magnetic stimulation (TMS) provides a non-invasive means for altering brain electrical neural activity. TMS sessions (sham/placebo and real TMS) will be conducted before two MRI scans with two weeks in-between to assess whether TMS stimulation to the visual cortex will enhance visual plasticity in patients with schizophrenia-spectrum disorders. This project may provide a better understanding of the underlying neurobiological mechanisms responsible for learning and memory deficits in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. age: 18-65,
2. no neurological illness, head trauma, or major medical illness,
3. not pregnant or nursing,
4. no contraindication for TMS or MRI scanning,
5. no current substance abuse/dependence.

Healthy controls will have no DSM-5 diagnosis and no first-degree relatives with a psychotic disorder.

Inclusion criteria for patients includes:

1. DSM-5 diagnosis of schizophreniform, schizophrenia or schizoaffective and competent to sign an informed consent,
2. not currently taking other medications that affects brain structure (e.g. steroids),
3. less than 12 months antipsychotic exposure and on the same psychotropic medications for 4 weeks prior to study,
4. not be taking clozapine (due to its effects on NMDA receptors and increase of seizure threshold),
5. clinically stable (i.e. no change in psychotic symptoms for at least 4 weeks).

Exclusion Criteria:

1. age outside of 18-65,
2. neurological illness, head trauma, or major medical illness,
3. pregnant or nursing,
4. contraindication for TMS or MRI scanning,
5. current substance abuse/dependence,
6. currently taking medications that affects brain structure (e.g. steroids).

Healthy controls with a DSM-5 diagnosis and/or a first-degree relative with a psychotic disorder. Participants with schizophrenia that are not competent to sign an informed consent, have more than 12 months antipsychotic exposure, not on the same psychotropic medications for 4 weeks prior to study, taking clozapine, and not clinically stable (i.e.a change in psychotic symptoms for at least 4 weeks).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Rowland, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 adults provided informed consent. 2 screen failures and 1 lost to follow-up before screening.
Groups:
- TMS (Active Then Sham): Participants first received active rTMS 10Hz to the occipital cortex and then 2 weeks later received sham (A sham coil was used to control for the auditory artifacts induced by rTMS)
  TMS: Transcranial Magnetic Stimulation
- TMS (Sham Then Active): Participants first received sham (A sham coil was used to control for the auditory artifacts induced by rTMS) and then 2 weeks later received active rTMS 10Hz to the occipital cortex
  TMS: Transcranial Magnetic Stimulation
- iTBS (Active Then Sham): Participants first received active iTBS 5 Hz to the occipital cortex and then 2 weeks later received sham (a sham coil was used to control for the auditory artifacts induced by iTBS).
  Intermittent theta-burst stimulation: iTBS
- iTBA (Sham Then Active): Participants first received sham (a sham coil was used to control for the auditory artifacts induced by iTBS) and then 2 weeks later received active iTBS 5 Hz to the occipital cortex .
  Intermittent theta-burst stimulation: iTBS
Period: Overall Study
Arm/Group | TMS (Active Then Sham) | TMS (Sham Then Active) | iTBS (Active Then Sham) | iTBA (Sham Then Active)
Started | 3 | 0 | 6 | 5
Completed | 3 | 0 | 5 | 5
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized to TMS (Sham then Active) condition
Groups:
- TMS (Active Then Sham): Participants first received active rTMS 10Hz to the occipital cortex and then 2 weeks later received sham (A sham coil was used to control for the auditory artifacts induced by rTMS)
- TMS (Sham Then Active): Participants first received sham (A sham coil was used to control for the auditory artifacts induced by rTMS) and then 2 weeks later received active rTMS 10Hz to the occipital cortex
- iTBS (Active Then Sham): Participants first received active iTBS 5 Hz to the occipital cortex and then 2 weeks later received sham (a sham coil was used to control for the auditory artifacts induced by iTBS).
- iTBS (Sham Then Active): Participants first received sham (a sham coil was used to control for the auditory artifacts induced by iTBS) and then 2 weeks later received active iTBS 5 Hz to the occipital cortex
- Total: Total of all reporting groups
Arm/Group | TMS (Active Then Sham) | TMS (Sham Then Active) | iTBS (Active Then Sham) | iTBS (Sham Then Active) | Total
Number analyzed (Participants) | 3 | 0 | 6 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 6 | 5 | 14
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (1) |  | 32.5 (10.6) | 33 (13.2) | 32.77 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 2 | 2 | 4
  Male | 3 |  | 4 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 0 | 0 | 1
  Not Hispanic or Latino | 2 |  | 6 | 5 | 13
  Unknown or Not Reported | 0 |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0 | 0
  Asian | 1 |  | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0
  Black or African American | 1 |  | 3 | 3 | 7
  White | 1 |  | 2 | 2 | 5
  More than one race | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 6 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: fMRI Blood Oxygenation Level Dependent (BOLD) Response of Visual Plasticity
Description: fMRI BOLD response in visual cortex, during visual stimulation (0.9 Hz) before and after high frequency visual stimulation (9 Hz).
Time Frame: ~1 hour
Population: 13 participants completed active and/or sham conditions for either TMS or iTBS
Measure: Mean (Standard Deviation); unit: Beta values
Groups:
- Patient: Active TMS 10 Hz: rTMS 10Hz to the occipital cortex
  TMS: Transcranial Magnetic Stimulation
- Patient: Sham TMS; Control: Sham TMS: A sham coil will be used. This condition controls for the auditory artifacts induced by rTMS.
  TMS: Transcranial Magnetic Stimulation
- Patient: Active iTBS; Control: Active iTBS: iTBS 5 Hz to the occipital cortex
  Intermittent theta-burst stimulation: iTBS
- Patient: Sham iTBS; Control: Sham iTBS: A sham coil will be used. This condition controls for the auditory artifacts induced by iTBS
  Intermittent theta-burst stimulation: iTBS
- Control: Active TMS 10 Hz: rTMS 10Hz to the occipital cortex
  Transcranial Magnetic Stimulation: Transcranial Magnetic Stimulation
Arm/Group | Patient: Active TMS 10 Hz | Patient: Sham TMS | Patient: Active iTBS | Patient: Sham iTBS | Control: Active TMS 10 Hz | Control: Sham TMS | Control: Active iTBS | Control: Sham iTBS
Number analyzed (Participants) | 1 | 1 | 7 | 6 | 2 | 2 | 3 | 3
Beta values | -2.95 (0) | -0.66 (0) | -0.29 (2.55) | 2.57 (4.17) | -0.7 (4.33) | 0.86 (2.33) | -2.44 (3.27) | 2.47 (1.36)

2. Secondary Outcome: Magnetic Resonance Spectroscopy (MRS) Assessment of Glutamate
Description: MRS was used to obtain occipital cortical glutamate levels (active, sham). Levels reflect institutional units, as is standard for the field.
Time Frame: ~1 hour
Population: 2 participants had missing data; 11 participants completed active and sham conditions for either TMS or iTBS
Measure: Mean (Standard Deviation); unit: spectroscopy institutional units
Arm/Group | Patient: Active TMS 10 Hz | Patient: Sham TMS | Patient: Active iTBS | Patient: Sham iTBS | Control: Active TMS 10 Hz | Control: Sham TMS | Control: Active iTBS | Control: Sham iTBS
Number analyzed (Participants) | 1 | 1 | 7 | 7 | 2 | 2 | 1 | 1
spectroscopy institutional units | 8.96 (NA) — sd cannot be computed on 1 person | 9.23 (NA) — sd cannot be computed on 1 person | 9.34 (1.19) | 9.16 (1.15) | 10.61 (0.49) | 9.97 (0.07) | 12.04 (NA) — sd cannot be computed on 1 person | 11.91 (NA) — sd cannot be computed on 1 person

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during active and sham sessions, 3 hours each, for up to 2 weeks.
Groups:
- Active TMS 10 Hz: rTMS 10Hz to the occipital cortex
  Transcranial Magnetic Stimulation: Transcranial Magnetic Stimulation
- Active iTBS: iTBS 5 Hz to the occipital cortex
  Intermittent theta-burst stimulation: iTBS
- Sham iTBS: A sham coil will be used. This condition controls for the auditory artifacts induced by iTBS
  Intermittent theta-burst stimulation: iTBS
Arm/Group | Active TMS 10 Hz | Sham TMS | Active iTBS | Sham iTBS
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers unable to statistically analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT03220438/Prot_SAP_001.pdf